CLINICAL TRIAL: NCT04287556
Title: Population at Risk of Malignant Hyperthermia: Ambispective Cohort.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: HUL-RHM-2019
Record Dates: First submitted 2020-02-04; First posted 2020-02-27 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-08

CONDITIONS: Hyperthermia, Malignant
MeSH Terms: conditions — Malignant Hyperthermia | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 50 variants have been described that can be considered "diagnostic mutations" of RYR1 and CACNA1S, and other under study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population in risk of MH: Patient with hypermetabolic response of skeletal musculature by causes related with Malignant Hyperthermia in the literature.
  Interventions: Diagnostic Test: In vitro contracture test (IVCT); Diagnostic Test: In vitro test of hypermetabolism in B lymphocytes; Diagnostic Test: Genetic test

INTERVENTIONS:
Diagnostic Test: In vitro contracture test (IVCT) — In vitro study of muscle contraction after exposure to different substances (caffeine and halothane).
Diagnostic Test: In vitro test of hypermetabolism in B lymphocytes — In vitro study of the activation of lymphocytes B after being incubated with a cocktail of primary antibodies and measuring the acidification in response to the RyR1, 4-CmC agonist, using ryanodine as a positive control.
Diagnostic Test: Genetic test — Analysis of genes related to MH (CACNA1S and RYR1).

SUMMARY:
Malignant hyperthermia (MH) is a pharmacogenetic disease that manifests itself as a hypermetabolic response of skeletal musculature, in genetically susceptible patients, with the inhalation of volatile halogenated anesthetics, depolarizing neuromuscular relaxants such and, rarely, physical stressors such as intense exercise and heat stroke.

HM diagnosis is based on the performance of two tests:

* In vitro muscle contraction test (IVCT): it is the gold standard of the diagnosis of HM in Europe.
* Pharmacogenetic study: about 50 genetic variants associated with HM have been described.

It also has been described that B lymphocytes of patients with MH have metabolic alterations.

The main objective is to evaluate the association of disorders that occur with hypermetabolic response of skeletal musculature and susceptibility to malignant hyperthermia (MH).

DETAILED DESCRIPTION:
Malignant hyperthermia (MH) is a pharmacogenetic disease that manifests itself as a hypermetabolic response of skeletal musculature, in genetically susceptible patients, with the inhalation of volatile halogenated anesthetics, depolarizing neuromuscular relaxants such and, rarely, physical stressors such as intense exercise and heat stroke.

Risk factors to present this disease are:

* An adverse reaction to general anesthesia manifested as an unexplained increase in carbon, dioxide production, tachycardia, temperature rise, muscle. stiffness, rhabdomyolysis, disseminated intravascular coagulation or death, or both. During anesthesia or within 60 minutes of treatment discontinuation.
* Family history of unexplained perioperative death.
* Postoperative rhabdomyolysis after clinical exclusion of other myopathies.
* Stress rhabdomyolysis, recurrent or persistent rhabdomyolysis increased serum creatine kinase concentration where no cause has been identified after neurological study (idiopathic hyperCKemia).
* Heat stroke by effort that requires hospital admission, where known predisposing factors have been excluded.
* Other myopaties Extreme physical activity, as well as environments with high temperatures favor the appearance of ischemia, anoxia and release of calcium from the sarcoplasmic reticulum, thus increasing the risk of developing MH.

There are also other infrequent diseases in which there is a ryanodine canalopathy by a mechanism similar to that seen in MH, but in cells of tissues other than skeletal striated muscle; as well as some drugs and other rare diseases that may be related to MH.

Despite the rarity of MH and given the severity of the disease clinic, it is mandatory to explore possible risks in patients with hypermetabolic response of skeletal musculature due to rare or trigger diseases (medications, drugs of abuse, exercise, extreme heat, others) whose MH risk is not defined.

Although the standard method for the diagnosis of MH is the in vitro test for halothane caffeine contraction (IVCT), it has been described that B lymphocytes of patients with MH have metabolic alterations. Alto, there are about 50 genetic variants associated with MH that have been described.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered at least one episode of rhabdomyolysis due to related causes in the literature with susceptibility to HM.
* Patients who have been given information about the study and have agreed to sign the consent of the study. The muscle biopsy will be performed under usual clinical practice.

Exclusion Criteria:

* Patients who have suffered episodes of rhabdomyolysis due to alternative causes: trauma, compression hypoxia during immobilization or loss of consciousness or infectious arterial occlusion (influenza A and B, coxackievirus, Epstein-Barr, HIV, legionella, Streptococcus pyogenes Staphilococcus aureus, clostridium), metabolic or electrolyte abnormalities (hypokalemia, hypophosphatemia, hypocalcemia, non-ketosic hyperosmolar conditions, diabetic ketoacidosis), others.
* Children under 10 years or less than 30 kg are excluded for the in vitro test (muscle biopsy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with hypermetabolic response of skeletal musculature by related causes in the literature with Malignant Hyperthermia.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Determination, by an in vitro study of muscular contraction, measuring the muscle tension, of the presence of Malignant Hyperthermia susceptibility in patients with a history of hypermetabolic response of skeletal musculature. | 5 years
  Measured by the tension induced by the muscular contraction in response to the presence of caffeine and halothane.
Determination, by genetic study, of the presence of susceptibility to Malignant Hyperthermia in patients with a history of hypermetabolic response of skeletal musculature. | 5 years
  Identifying determined genes related with Malignant Hyperthermia risk.
Study of the concordance of the genetic study and IVCT versus the hypermetabolic response of B lymphocyte, in patients with a history of hypermetabolic response of skeletal musculature. | 5 years
  Extracellular acidification curve in B lymphocytes in response to the agonist RyR1 and 4-CmC.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ramírez García, Principal Investigator — Clinical Pharmacology Department, La Paz University Hospital
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain